CLINICAL TRIAL: NCT02169362
Title: Phase I, Double-Blind, Randomized, Controlled Study to Demonstrate the Safety of Applying Autologous Platelet Rich Plasma (PRP) Gel (Magellan® Bio-Bandage™) to Acute Deep Partial Thickness Thermal Injuries
Brief Title: Applying Platelet Rich Plasma (PRP) Gel to Acute Deep Partial Thickness Thermal Injuries
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Arteriocyte, Inc. (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: ART 13-005; IDE 15921 (Other: Center for Biologics Evaluation and Research)
Record Dates: First submitted 2014-05-23; First posted 2014-06-23 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-01

CONDITIONS: Acute Deep Partial Thickness Thermal Burns
Keywords: Burns; Thermal burns; Second degree burns; Partial thickness burns; Deep partial thickness burns; Acute burns; Burn wounds
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Platelet Rich Plasma - Bio-Bandage™ (Experimental): Autologous Platelet Rich Plasma (PRP) Gel (Magellan® Bio-Bandage™)
  Interventions: Device: Autologous Platelet Rich Plasma (PRP) Gel (Magellan® Bio-Bandage™)
- Saline Spray, Standard of Care (Sham Comparator)
  Interventions: Device: Autologous Platelet Rich Plasma (PRP) Gel (Magellan® Bio-Bandage™)

INTERVENTIONS:
Device: Autologous Platelet Rich Plasma (PRP) Gel (Magellan® Bio-Bandage™) — Application of up to 18 mL of autologous PRP gel (Magellan® Bio-Bandage™) to the surface of an acute deep partial thickness burn wound no greater than 72 cm squared within 72 hours of the initial injury. Intervention is in addition to standard of care treatment. The PRP Bio-Bandage™ is prepared using the Magellan® System and is FDA cleared via BK030040 and BK040068.
  Other Names: The Magellan® System

SUMMARY:
The study will examine the safety of using a concentration of proteins from a patient's own blood, referred to as platelet rich plasma or (PRP) and applying it to a second degree burn wound.

DETAILED DESCRIPTION:
The objective of this trial is to demonstrate the safety of applying autologous PRP gel (Magellan® Bio-Bandage™) to acute deep partial thickness thermal burns in the first days after burn injury.

The Magellan® Bio-Bandage™ Burn Wound Care Kit is intended for the preparation and application of an autologous biological covering to deep partial thickness burn wounds to delay or minimize skin grafting requirements.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent will be obtained prior to study participation
* Male or female age ≥ 18 years of age or ≤ 86 years of age
* Total burn wound measuring ≤ 25% TBSA
* Burn wound area to be treated must be a deep partial thickness wound
* Burn wound area to be treated must be ≤72 cm2 and surrounded by a perimeter of healthy skin
* Able and willing to comply with the procedures required by the protocol. Subjects may be managed as either inpatient or outpatient.
* If a female of childbearing potential, the subject must have a negative serum pregnancy test at screening
* All subjects, male and female, must use acceptable method(s) of birth control for the duration of the study
* Female subjects must be of non childbearing potential (defined as postmenopausal for at least 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy or hysterectomy]) or must be using adequate contraception (practicing one of the following methods of birth control):
* Total abstinence from sexual intercourse (minimum of one complete menstrual cycle before study entry)
* A partner who is physically unable to impregnate the subject (e.g., vasectomized)
* Contraceptives (oral, parenteral, or transdermal) for 3 consecutive months prior to subject's cell concentrate administration
* Intrauterine device (IUD), or
* Double barrier method (condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream)

Exclusion Criteria:

* Conductive electrical, friction or chemical burns
* Burns to the digits, head, genitalia, palms of hands, soles of feet, and face that are the only possible sites for treatment (subjects with burns elsewhere in addition to these sites may be enrolled in the study)
* Burns that pose a risk to digits or limbs
* Subjects who have gone into hemorrhagic shock following burn injury
* Subject was medically treated for insulin-dependent or non-insulin-dependent diabetes mellitus prior to burn injury per subject medical history
* Venous or arterial vascular disorder directly affecting a designated test area
* Known immune deficiency disorder, either congenital or acquired
* Chronically malnourished as determined clinically by the investigator. (Investigators are responsible for determining if subjects are chronically malnourished during the screening process. Investigators should take into consideration the following parameters: medical history and physical appearance, the subject's body mass index, and any significant laboratory findings)
* Severe respiratory problems or concurrent head trauma at hospital admission, including inhalation injury requiring ventilator support
* Any chronic condition requiring the use of systemic corticosteroids 30 days prior to study entry and anytime during the course of the study
* Use of COX-1 and/or COX-2 inhibitors within 48 hours prior to treatment. Subjects must refrain from use of NSAIDs for five days after Visit 2.
* Any other acute or chronic concurrent medical condition(s) that, in the investigator's opinion, are a contraindication to study participation or limit the subject's life expectancy to < 6 months
* Known or suspected hypersensitivity to Recothrom®
* Concurrent participation in another clinical trial in which an investigational agent is used. (Subjects must not have been enrolled in another clinical trial within 30 days of enrolling in this trial)
* Females who are pregnant or nursing or intend to become pregnant during the duration of the study
* Burn wounds that occur over joints
* Known allergies to silver, adhesive products or silicone.
* Subjects with the following abnormal laboratory test levels:
* Stage 4 or greater chronic kidney disease (eGFR < 30 mL/min
* Hemoglobin < 10 g/dl
* Thrombocytopenia < 100,000 platelets/µl.
* Serum albumin level < 2.5 g/dl or > 30 g/dl at time of screening
* Liver function*:
* AST- Males and Females, >2.5 ULN
* ALT- Males and Females, >2.5 ULN
* Alkaline Phosphatase- Males and Females: >2.0 ULN
* Total bilirubin- Males and Females >2.0 ULN

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-07; Primary Completion 2018-01 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by Adverse Events | Days 1 -365
  The primary objective of this trial is to demonstrate the safety of applying autologous PRP gel to acute deep partial thickness thermal burns in the first days after burn injury. The primary endpoint of this study will be safety. Incidence of Adverse Events and/or Serious Adverse Events will be documented, along with time to wound closure.

SECONDARY OUTCOMES:
Delay or minimization of skin grafting requirements following burn injury | Change will be assessed up to 35 Days
  This outcome will be evaluated by time to graft (days), need for graft (yes or no), and incidence of graft occurrence ( percentage of subjects in control group versus treatment group requiring a skin graft).
Improved wound healing trajectory as compared to standard of care | Change will be assessed up to 365 Days
  Wound healing will be assessed by calculating wound size measurements and percentage of change over time utilizing digital photography and planimetry software.
Increased rate of wound closure as compared to standard of care | Change will be assessed up to 365 Days
  The percentage of treated subjects versus standard of care only subjects with complete wound closure at 28 and 42 days post-burn injury. Wound closure will be defined as skin re-epithelialization without drainage or dressing requirements confirmed at two consecutive visits.
Reduced scarring, pain and pruritus | Change will be assessed up to 365 Days
  This outcome will compare treated subjects to standard of care only subjects by analyzing photo images and scar scale analysis (principal investigator and blinded rater assessments), and based on subject reported pain and pruritus.
Improved Skin-Healing Quality | Change will be assessed up to 365 Days
  Histological analysis of 2mm skin biopsies taken at Baseline (Day 1) and 90 days post-treatment will be analyzed and compared. Biopsies will be taken only from subject for whom a skin graft was not required, and from both treated subjects and standard of care only subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Barnes, PhD, Study Director — Arteriocyte, Inc.
Locations (8):
- United States (8):
  - Arizona Burn Center, Phoenix, Arizona
  - University of California, Davis Medica Center, Sacramento, California
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - Tampa General Hospital/University of South Florida, Tampa, Florida
  - University Medical Center Southern Nevada, Lions Regional Burn Center, Las Vegas, Nevada
  - Jaycee Burn Center at University of North Carolina, Chapel Hill, North Carolina
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - Firefighters' Regional Burn Center, Memphis, Tennessee

REFERENCES:
- [Background] Badiavas AR, Badiavas EV. Potential benefits of allogeneic bone marrow mesenchymal stem cells for wound healing. Expert Opin Biol Ther. 2011 Nov;11(11):1447-54. doi: 10.1517/14712598.2011.606212. Epub 2011 Aug 20. PMID 21854302
- [Background] Barr JE. Principles of wound cleansing. Ostomy Wound Manage. 1995 Aug;41(7A Suppl):15S-21S; discussion 22S. PMID 7669196
- [Background] Almdahl SM, Veel T, Halvorsen P, Vold MB, Molstad P. Randomized prospective trial of saphenous vein harvest site infection after wound closure with and without topical application of autologous platelet-rich plasma. Eur J Cardiothorac Surg. 2011 Jan;39(1):44-8. doi: 10.1016/j.ejcts.2010.06.007. Epub 2010 Jul 15. PMID 20634084
- [Background] Bielecki TM, Gazdzik TS, Arendt J, Szczepanski T, Krol W, Wielkoszynski T. Antibacterial effect of autologous platelet gel enriched with growth factors and other active substances: an in vitro study. J Bone Joint Surg Br. 2007 Mar;89(3):417-20. doi: 10.1302/0301-620X.89B3.18491. PMID 17356164
- [Background] Boswell SG, Cole BJ, Sundman EA, Karas V, Fortier LA. Platelet-rich plasma: a milieu of bioactive factors. Arthroscopy. 2012 Mar;28(3):429-39. doi: 10.1016/j.arthro.2011.10.018. Epub 2012 Jan 28. PMID 22284405
- [Background] Bush J, Duncan JAL, Bond JS, Durani P, So K, Mason T, O'Kane S, Ferguson MWJ. Scar-improving efficacy of avotermin administered into the wound margins of skin incisions as evaluated by a randomized, double-blind, placebo-controlled, phase II clinical trial. Plast Reconstr Surg. 2010 Nov;126(5):1604-1615. doi: 10.1097/PRS.0b013e3181ef8e66. PMID 21042116
- [Background] Church D, Elsayed S, Reid O, Winston B, Lindsay R. Burn wound infections. Clin Microbiol Rev. 2006 Apr;19(2):403-34. doi: 10.1128/CMR.19.2.403-434.2006. PMID 16614255
- [Background] Dib N, Michler RE, Pagani FD, Wright S, Kereiakes DJ, Lengerich R, Binkley P, Buchele D, Anand I, Swingen C, Di Carli MF, Thomas JD, Jaber WA, Opie SR, Campbell A, McCarthy P, Yeager M, Dilsizian V, Griffith BP, Korn R, Kreuger SK, Ghazoul M, MacLellan WR, Fonarow G, Eisen HJ, Dinsmore J, Diethrich E. Safety and feasibility of autologous myoblast transplantation in patients with ischemic cardiomyopathy: four-year follow-up. Circulation. 2005 Sep 20;112(12):1748-55. doi: 10.1161/CIRCULATIONAHA.105.547810. PMID 16172284
- [Background] Erbs S, Linke A, Adams V, Lenk K, Thiele H, Diederich KW, Emmrich F, Kluge R, Kendziorra K, Sabri O, Schuler G, Hambrecht R. Transplantation of blood-derived progenitor cells after recanalization of chronic coronary artery occlusion: first randomized and placebo-controlled study. Circ Res. 2005 Oct 14;97(8):756-62. doi: 10.1161/01.RES.0000185811.71306.8b. Epub 2005 Sep 8. PMID 16151021
- [Background] Farrior E, Ladner K. Platelet gels and hemostasis in facial plastic surgery. Facial Plast Surg. 2011 Aug;27(4):308-14. doi: 10.1055/s-0031-1283050. Epub 2011 Jul 26. PMID 21792775
- [Background] Fearmonti R, Bond J, Erdmann D, Levinson H. A review of scar scales and scar measuring devices. Eplasty. 2010 Jun 21;10:e43. PMID 20596233
- [Background] Fearmonti RM, Bond JE, Erdmann D, Levin LS, Pizzo SV, Levinson H. The modified Patient and Observer Scar Assessment Scale: a novel approach to defining pathologic and nonpathologic scarring. Plast Reconstr Surg. 2011 Jan;127(1):242-247. doi: 10.1097/PRS.0b013e3181f959e8. PMID 21200219
- [Background] Forrester JS, Price MJ, Makkar RR. Stem cell repair of infarcted myocardium: an overview for clinicians. Circulation. 2003 Sep 2;108(9):1139-45. doi: 10.1161/01.CIR.0000085305.82019.65. No abstract available. PMID 12952828
- [Background] Gunaydin S, McCusker K, Sari T, Onur M, Gurpinar A, Sevim H, Atasoy P, Yorgancioglu C, Zorlutuna Y. Clinical impact and biomaterial evaluation of autologous platelet gel in cardiac surgery. Perfusion. 2008 May;23(3):179-86. doi: 10.1177/0267659108097783. PMID 19029269
- [Background] Jorgensen B, Karlsmark T, Vogensen H, Haase L, Lundquist R. A pilot study to evaluate the safety and clinical performance of Leucopatch, an autologous, additive-free, platelet-rich fibrin for the treatment of recalcitrant chronic wounds. Int J Low Extrem Wounds. 2011 Dec;10(4):218-23. doi: 10.1177/1534734611426755. Epub 2011 Oct 18. PMID 22009148
- [Background] Kazakos K, Lyras DN, Verettas D, Tilkeridis K, Tryfonidis M. The use of autologous PRP gel as an aid in the management of acute trauma wounds. Injury. 2009 Aug;40(8):801-5. doi: 10.1016/j.injury.2008.05.002. Epub 2008 Aug 13. PMID 18703188
- [Background] Keck M, Selig HF, Lumenta DB, Kamolz LP, Mittlbock M, Frey M. The use of Suprathel((R)) in deep dermal burns: first results of a prospective study. Burns. 2012 May;38(3):388-95. doi: 10.1016/j.burns.2011.09.026. Epub 2011 Nov 10. PMID 22078803
- [Background] Khalafi RS, Bradford DW, Wilson MG. Topical application of autologous blood products during surgical closure following a coronary artery bypass graft. Eur J Cardiothorac Surg. 2008 Aug;34(2):360-4. doi: 10.1016/j.ejcts.2008.04.026. Epub 2008 Jun 26. PMID 18585051
- [Background] Lee H. Outcomes of sprayed cultured epithelial autografts for full-thickness wounds: a single-centre experience. Burns. 2012 Sep;38(6):931-6. doi: 10.1016/j.burns.2012.01.014. Epub 2012 Jun 9. PMID 22688194
- [Background] Saad Setta H, Elshahat A, Elsherbiny K, Massoud K, Safe I. Platelet-rich plasma versus platelet-poor plasma in the management of chronic diabetic foot ulcers: a comparative study. Int Wound J. 2011 Jun;8(3):307-12. doi: 10.1111/j.1742-481X.2011.00797.x. Epub 2011 Apr 7. PMID 21470370
- [Background] Schwacha MG, Nickel E, Daniel T. Burn injury-induced alterations in wound inflammation and healing are associated with suppressed hypoxia inducible factor-1alpha expression. Mol Med. 2008 Sep-Oct;14(9-10):628-33. doi: 10.2119/2008-00069.Schwacha. PMID 18615157
- [Background] Serraino GF, Dominijanni A, Jiritano F, Rossi M, Cuda A, Caroleo S, Brescia A, Renzulli A. Platelet-rich plasma inside the sternotomy wound reduces the incidence of sternal wound infections. Int Wound J. 2015 Jun;12(3):260-4. doi: 10.1111/iwj.12087. Epub 2013 May 21. PMID 23692143
- [Background] Sullivan T, Smith J, Kermode J, McIver E, Courtemanche DJ. Rating the burn scar. J Burn Care Rehabil. 1990 May-Jun;11(3):256-60. doi: 10.1097/00004630-199005000-00014. PMID 2373734
- [Background] Trowbridge CC, Stammers AH, Woods E, Yen BR, Klayman M, Gilbert C. Use of platelet gel and its effects on infection in cardiac surgery. J Extra Corpor Technol. 2005 Dec;37(4):381-6. PMID 16524157
- [Background] Valeri CR, Saleem B, Ragno G. Release of platelet-derived growth factors and proliferation of fibroblasts in the releasates from platelets stored in the liquid state at 22 degrees C after stimulation with agonists. Transfusion. 2006 Feb;46(2):225-9. doi: 10.1111/j.1537-2995.2006.00705.x. PMID 16441599
- [Background] Wolf SE, Arnoldo BD. The year in burns 2012. Burns. 2013 Dec;39(8):1501-13. doi: 10.1016/j.burns.2013.11.001. Epub 2013 Nov 16. PMID 24252249